CLINICAL TRIAL: NCT05982899
Title: A Web-based Calculator Predicts Heterogeneous Frailty Trajectories Among Elderly Gastric Cancer Survivors
Brief Title: A Web-based Calculator Predicts Heterogeneous Frailty Trajectories
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xueyi Miao, Principal Investigator, Nanjing Medical University
Other Study IDs: 2020-273
Record Dates: First submitted 2023-07-22; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Gastric Cancer
Keywords: gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the predictive factors of frailty trajectories and develop a web-based nomogram among gastric cancer survivors.

DETAILED DESCRIPTION:
The aims of this study are to explore the predictive factors of frailty trajectories in gastric cancer patients more comprehensively based on the health ecology theory and to construct a clinically convenient web-based prediction calculator, so as to screen high-risk frailty elderly gastric cancer patients at an early stage in clinical practice, and thus to implement early interventions to improve the prognosis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with gastric cancer by endoscopy or pathology;
* age ≥60 years old;
* radical gastrectomy was proposed;
* be able to communicate simply in writing and verbally.

Exclusion Criteria:

* combined with other sites of malignant tumors;
* combined with severe heart, liver, lung, and renal insufficiency;
* recent using hormones, immunosuppressants;
* with physical disabilities.

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: elderly gastric cancer survivors
Sampling Method: Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
frailty trajectories | 1 year
  Frailty was measured by Tilburg frailty indicator (TFI) scale at discharge, one month, three months, six months and twelve months after surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xueyi Miao, Nanjing, Jiangsu
  - Nanjing medical university, Nanjing

REFERENCES:
- [Derived] Guo Y, Miao X, Chen Y, Ding L, Zhao K, Xu T, Chen L, Xu X, Xu Q. Hypothetical Interventions on Frailty Heterogeneous Trajectories of Older Patients with Gastric Cancer Using Parametric G-Formula. Ann Surg Oncol. 2025 Oct;32(10):7634-7643. doi: 10.1245/s10434-025-18026-w. Epub 2025 Aug 9. PMID 40783664
- [Derived] Miao X, Guo Y, Ding L, Xu X, Zhao K, Zhu H, Chen L, Chen Y, Zhu S, Xu Q. A dynamic online nomogram for predicting the heterogeneity trajectories of frailty among elderly gastric cancer survivors. Int J Nurs Stud. 2024 May;153:104716. doi: 10.1016/j.ijnurstu.2024.104716. Epub 2024 Feb 13. PMID 38412776